CLINICAL TRIAL: NCT01104922
Title: Re-irradiation With Fractionated Stereotactic Radiosurgery Plus Cetuximab in Patients With Recurrent Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David A. Clump, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, David A. Clump, MD, PhD, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 06-093
Record Dates: First submitted 2010-04-08; First posted 2010-04-16 (Estimated); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Fractionated Stereotactic Radiosurgery
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cetuximab and stereotactic radiosurgery (Experimental)
  Interventions: Drug: Cetuximab; Device: Stereotactic radiosurgery

INTERVENTIONS:
Drug: Cetuximab — Cetuximab will be administered for 3 weekly doses commencing one week prior to stereotactic radiosurgery treatment as follows: * Cetuximab 400 mg / m2 day -7 (1 week prior to initiation of radiosurgery) * Cetuximab 250 mg/m2 days 0 and +8 (i.e. during the first and second week of fractionated stereotactic radiosurgery) Cetuximab will be administered at 400 mg/m2 IV over 120 minutes on day -7 (loading dose) and 250 mg/m2 IV on days 0 and 8 during the course of stereotactic radiosurgery.
  Other Names: Erbitux
Device: Stereotactic radiosurgery — Fractionated stereotactic radiosurgery, 8.0 Gy per fraction for 5 fractions (total: 40.0 Gy)

SUMMARY:
This trial examines survival and toxicity in previously irradiated patients with squamous cell carcinoma of the head and neck (SCCHN) treated with radiosurgery and cetuximab and to evaluate the acute and late toxicities associated with the above therapy.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the head and neck is the sixth most common malignancy worldwide with approximately 500,000 cases worldwide yearly. There were an estimated 39,250 new cases and 11,000 deaths in the United States in 2005 (Jemal 2005, Spitz MR). Despite major improvements in the treatment of SCCHN in recent years which include the introduction of concurrent chemoradiotherapy as an effective primary or postoperative therapy, the five-year survival rate for patients with SCCHN in the United States and other developed countries remains poor as nearly 50-60% of these patients will die as a direct result of recurrent locoregional disease. This study aims to determine the 1-year progression-free survival (PFS) of previously irradiated patients with squamous cell carcinoma of the head and neck (SCCHN) treated with radiosurgery and cetuximab and to evaluate the acute and late toxicities associated with the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven recurrent squamous cell carcinoma of the head and neck (SCCHN), who has received prior radiotherapy with or without chemotherapy. New primary is allowed if location is in a previously irradiated field. Biopsy is recommended for each recurrence; but is not mandated per study. This will be at the discretion of the principal investigator.
* Prior radiation dose of at least 60 Gy.
* Disease confined to locoregional site and can be encompassed in a stereotactic radiosurgery "portal"
* Tumor must be deemed to be inoperable or unresectable either by clinical or radiographic criteria. These criteria include encasement of great vessels, vertebral invasion or undue peri-operative risk.
* Prior surgery for recurrent or new SCCHN is allowed in previously irradiated patients. A minimum of 4 weeks should elapse between any surgery and treatment on study. However, high risk pathologic features should be present, such as positive margins, positive lymphadenopathy, perineural or angiolymphatic invasion. Measurable disease must be present for assessment of response.
* Karnofsky performance status > 60 (ECOG 0-2)
* Prior treatment with an EGFR Inhibitor is allowed if it was a part of prior curative therapy and was completed at least 30 days prior to commencement of study therapy
* Any number of prior chemotherapy regimens are allowed
* Measurable disease on imaging studies (MRI, CT, PET-CT or physical exam)
* Age > 18
* Estimated life expectancy > 12 weeks
* No prior radiation therapy or chemotherapy within 1 month of study enrollment
* No prior chemotherapy or targeted therapy within the previous 4 weeks
* ANC > 1000, PLT>75,000, Serum creatinine<2.5 mg/dL, Bilirubin <1.5 x upper limits of normal (ULN)
* Diabetes must be controlled prior to PET-CT scanning (blood glucose <200 mg/dL)
* Ability to provide written informed consent

Exclusion Criteria:

* Evidence of distant metastasis on upright chest x-ray (CXR), computed tomography (CT) or other staging studies
* History of any cancer other than SCCHN (except non-melanoma skin cancer or carcinoma in situ of the cervix) within the last 5 years.
* Patients in their reproductive age group should use an effective method of birth control. Patients who are breast-feeding, or have a positive pregnancy test will be excluded from the study
* Any co-morbidity or condition of sufficient severity to limit full compliance with the protocol per assessment by the investigator
* Concurrent serious infection
* History of known hypersensitivity to cetuximab or similar agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-12-26 (Actual); Primary Completion 2014-05-21 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Clump, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vargo JA, Ferris RL, Ohr J, Clump DA, Davis KS, Duvvuri U, Kim S, Johnson JT, Bauman JE, Gibson MK, Branstetter BF, Heron DE. A prospective phase 2 trial of reirradiation with stereotactic body radiation therapy plus cetuximab in patients with previously irradiated recurrent squamous cell carcinoma of the head and neck. Int J Radiat Oncol Biol Phys. 2015 Mar 1;91(3):480-8. doi: 10.1016/j.ijrobp.2014.11.023. Epub 2015 Jan 30. PMID 25680594

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Prior surgery [Number; unit: percentage of participants] | 67
Prior chemotherapy [Number; unit: percentage of participants] | 65
Received prior epidermal growth factor receptor (EGFR) [Number; unit: percentage of participants] | 23
Zubrod performance status [Count of Participants; unit: Participants] — A scale for indicating a patient's functional level: 0 asymptomatic - 1 Symptomatic, fully ambulatory - 2 Symptomatic, in bed - 50% of the day - 3 Symptomatic, in bed > 50% of the day but not bedridden - 4 Bedridden - 5 Dead.
  Participants
    Score = 0 | 22
    Score = 1 | 23
    Score = 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: 1-year Local Progression-free Survival (PFS)
Description: Progression (response as assessed by subjective interpretation of the first PET-CT) per Response Evaluation Criteria in Solid Tumors (RECIST v1.0) was defined as greater than 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum and longest diameter recorded since the baseline measurements or the appearance of 1 or more new lesion(s). If the measurable disease was restricted to a solitary lesion, the protocol specified that neoplastic nature should be confirmed by cytology and histology.
Time Frame: At 1-year
Population: Patients that received study therapy and were evaluable for response to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Number analyzed (Participants) | 48
percentage of participants | 60 [44 to 75]

2. Primary Outcome: 1-year Locoregional Progression-free Survival (PFS)
Description: as for outcome 1
Time Frame: At 1-year
Population: Patients that received study therapy and were evaluable for response to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Number analyzed (Participants) | 48
percentage of participants | 37 [23 to 53]

3. Primary Outcome: 1-year Distant Progression-free Survival (PFS)
Description: as for outcome 1
Time Frame: At 1-year
Population: Patients that received study therapy and were evaluable for response to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Number analyzed (Participants) | 48
percentage of participants | 77 [54 to 85]

4. Secondary Outcome: 1-year Progression-free Survival (PFS)
Description: Progression was defined as greater than 20% increase in the sum of the longest diameters of target lesions, per Response Evaluation Criteria in Solid Tumors (RECIST v1.0), taking as reference the smallest sum and longest diameter recorded since the baseline measurements or the appearance of 1 or more new lesion(s). If the measurable disease was restricted to a solitary lesion, the protocol specified that neoplastic nature should be confirmed by cytology and histology.
Time Frame: At 1-year
Population: Patients that received study therapy and were evaluable for response to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Number analyzed (Participants) | 48
percentage of participants | 33 [20 to 49]

5. Secondary Outcome: Overall Survival (OS)
Description: Number of months patients remaining alive after study treatment.
Time Frame: Up to 2 years
Population: Patients that received study therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Number analyzed (Participants) | 48
months | 10 [7 to 16]

6. Secondary Outcome: Overall Response (OR)
Description: Response by number and percentage of patients assessed by subjective interpretation of the first PET-CT. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response(CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Up to 2 years
Population: Patients that received study therapy and were evaluable for response to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Number analyzed (Participants) | 48
Participants
  Complete response | 9
  Partial Response | 13
  Stable disease | 5
  Disease progression | 17

7. Secondary Outcome: Changes in Tumor Glucose Metabolism
Description: Glucose metabolism was assessed by FDG PET. FDG uptake reflects the tissue glucose metabolism and is usually high in high-grade tumors and relatively low in low-grade tumors.
Time Frame: Up to 24 months / post therapy
Population: Patients that received study therapy and were evaluable for response and by FDG PET.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Number analyzed (Participants) | 44
Participants
  Complete Response (CR) | 9
  Partial Response (PR) | 13
  Stable Disease (SD) | 5
  Progressive Disease (PD) | 17

8. Secondary Outcome: Changes in Tumor Hypoxia.
Description: Changes in tumor hypoxia (tumor cells deprived of oxygen) as a result of Stereotactic radiosurgery (SRS) through assessment by pre-and post-treatment fluorodeoxyglucose (FDG)- and fluoromisonidazole (FMISO)-PET.
Time Frame: Up to 24 months; before and after treatment
Population: At the time of this study, PMISO could not be readily obtained due to its relatively short half-life and unforeseen inability to procure this radioisotope locally. Thus, to prevent delay in treating aggressive cancer, F-MISO scans were not performed.
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Number analyzed (Participants) | 0

9. Secondary Outcome: Quality of Life (QoL)
Description: Percentage of patients that reported stable and/or improved of quality of life after SBRT as indicated by a quantitative increase or maintenance in overall score. Quality of Life was assessed by longitudinal collection of the University of Washington Quality of Life Registry (UW-QoL-R) survey data, both pre- and post-SBRT. Patients completed the previously validated UW-QoL-R survey at enrollment and again after SBRT. UW-QoL-R measures patient reported QoL in 12 head and neck-specific and 3 global health domains, using a single Likert-scale question with an assigned score of 0 to 100 with 100 representing normal function.
Time Frame: Baseline, 6-8 weeks post-treatment; up to 16 months
Population: Patients that received study therapy and were able to complete Quality of Life assessments, who reported stable or improved quality of life.
Measure: Number; unit: percentage of participants
Arm/Group | Cetuximab and Stereotactic Radiosurgery
Number analyzed (Participants) | 28
percentage of participants | 62

ADVERSE EVENTS:
Time Frame: Adverse events were assessed through study completion, up to 2 years.
Description: Adverse Events and Serious Adverse Events determined using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 Adverse Events were Grade 1 and Grade2 toxicities; Serious Adverse Events were Grade 3 and Grade 4 toxicities.
  All-Cause Mortality: At last follow-up, 69% died of disease, 4% died with disease, 15% died without progression, 10% were alive without progression, and 2% were alive with progression; 88% deceased at time of final analysis.
Arm/Group | Cetuximab and Stereotactic Radiosurgery
All-Cause Mortality (participants affected / at risk) | 42/48
Serious Adverse Events (participants affected / at risk) | 3/48
Other Adverse Events (participants affected / at risk) | 43/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab and Stereotactic Radiosurgery (N=48)
Dysphagia (Gastrointestinal disorders) | 1
Rash (erbiutx) (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab and Stereotactic Radiosurgery (N=48)
Dry Mouth (Xerostomia) (Gastrointestinal disorders) | 8
Dysgeusia (Taste Alteration (Gastrointestinal disorders) | 4
Mucositis (Gastrointestinal disorders) | 26
Dysphagia (Gastrointestinal disorders) | 9
Odynphagia (Painful swallowing) (Gastrointestinal disorders) | 8
Dysphonia (difficulty speaking) (Gastrointestinal disorders) | 1
Voice Changes (hoarsenss) (Respiratory, thoracic and mediastinal disorders) | 2
Pain (General disorders) | 5
Fatigue (General disorders) | 5
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Rash (erbiutx) (Skin and subcutaneous tissue disorders) | 15
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 6
Fibrosis (Skin and subcutaneous tissue disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes